CLINICAL TRIAL: NCT06994754
Title: Evaluation of Maxillary Expansion Using Clear Aligners' Therapy in Patients With Cleft Lip and Palate at the Mixed Dentition Stage: A Pilot Study
Brief Title: Evaluation of Maxillary Expansion Using Clear Aligners' Therapy in Patients With Cleft Lip and Palate at the Mixed Dentition Stage
Acronym: Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mahmoud abdelsalam, Master degree candidate at Orthodontic Department, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTH 3-3-7
Record Dates: First submitted 2025-03-29; First posted 2025-05-29 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Maxillary Deficiency; Cleft Lip and Palate
Keywords: Maxillary Expansion by Aligners
MeSH Terms: conditions — Retrognathia; Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bilateral cleft lip and palate patients (Experimental)
  Interventions: Device: clear aligners

INTERVENTIONS:
Device: clear aligners — aligners made with 1mm thickness sheet and covering the whole palate

SUMMARY:
The goal of this clinical trial is to learn if the aligners can expand upper dental arch in patients with cleft lip and palate at age of 6-8 years old to correct their collapsid archs. The main questions it aims to answer are:

Does aligners can achieve transverse dento-skeletal changes? Does aligners can achieve anteroposterior and vertical dento-skeletal changes?

Participants will:

Wear sequence of aligners (each for 10 days). Visit the clinic every month for checkups. 3D x-ray and intraoral scan will be taken after completion of the aligners set to evaluate the intervention.

DETAILED DESCRIPTION:
Cleft lip and palate (CLP) is the most prevalent among all craniofacial anomalies, affecting one in every 700 births and disturbing the quality of life of more than 7 million people around the world.

Cleft lip and palate are defined as malformations characterized by the non-union of the upper lip and/or palate, either separately or in conjunction with another syndrome. Its etiology is rather complex and definitely multifactorial, where complex interplay between genetic and environmental factors play a significant role in the incidence and cause of cleft.

Cleft lips can be unilateral or bilateral, and may involve the alveolus or palate. Unilateral cleft lip shows a 2:1 left predominance.

Lip and palate surgical repairs are performed in the first months and years of life respectively. As a consequence, the growth and development of the maxillary segments are compromised by scar tissues, presenting a significant maxillary transverse deficiency with medially collapsed cleft segments accompanied with anterior crossbite or both anterior and posterior crossbites. Most CLP patients present a narrower anterior than posterior maxillary arch frequently showing a crossbite in both canine and premolar areas and a normal occlusal transverse molar relationship.

Maxillary expansion is usually performed before the secondary alveolar bone grafting procedure. Expansion improves the maxillary arch morphology and causes the segmental alignment creating appropriate conditions for bone grafting surgery as well as correcting the posterior crossbites.

Variable appliances have been used for maxillary arch expansion in cleft patients for example Quad-helix, Hyrax and Haas expanders with its modifications with or without teeth alignment.

The investigators will conducted this clinical trial to evaluate if clear aligners (the new substitute to the conventional metal orthodontics) can achieve true dentoskeletal expansion in the three dimensions.

After clinical examination, intraoral scan taken also intra-oral and extra-oral photos. Requesting full skull CBCT.

Segmentation of teeth and palate using 3-shape software. Using aligner module to plan around 8-12 aligners with maximum velocity of 0.3 mm translation and 3 degree of rotation.

Exporting the models and fabrication of aligners using 1 mm thickness sheets. Delivery of aligners to the patient. Follow up every month. Full face CBCT and intraoral scan will be taken after completion of the intervention.

Measuring and superimpose the data before and after to extract the results.

ELIGIBILITY:
Inclusion Criteria:

* Mixed dentition.
* Both males and females.
* Bilateral cleft lip and palate.
* Lip repair performed between 3 and 6 months of age and palate repair performed between 12and 24 months of age.
* Presence of maxillary constriction that needs maxillary expansion.
* Good periodontal health.
* No previous orthodontic treatment.

Exclusion Criteria:

* Syndromic cleft lip and palate patients.
* Taking medications that influence growth.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Transverse dento-skeletal changes | six months
  Using pre and post treatment cone beam computed tomography (CBCT), 3D point identification and landmark development will be done. On the CBCT, skeletal transvers maxillary width, anterior, middle and posterior cleft width, intermolar, inter premolar and inter-canine widths will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Cairo University, Cairo, Select, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial